CLINICAL TRIAL: NCT03324217
Title: Effects of Motor Imagery and Action Observation on Electromyographic Activity and Intramuscular Oxygenation in the Hand Gripping Gesture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: uamadrid 3
Record Dates: First submitted 2017-10-20; First posted 2017-10-27 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Asymptomatic Subjects; Painfree Voluntiers; Neuroscience
Keywords: motor imagery; action observation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Imagery Group (Experimental): The participants in the motor imagery group were given instructions to perform a daily training composed of two sets of activities. The main set consisted of 10 isometric hand grip contractions for 3 seconds each with a tennis ball, leaving a 20-second break between contractions. In the first set, the participant only had to imagine that he was performing that task, placed in the standard position with the tennis ball in the hand. Once the first set was completed, the participant had to take a 2-minute break before starting the second set, in which they had to complete the set both imagining and actively performing the isometric contractions with the tennis ball.
  Interventions: Other: Mental Practise
- Action Observation Group (Experimental): The participants in the action observation group were given instructions to perform a daily training comprised of two sets of activities. The main set consisted of 10 isometric hand grip contractions for 3 seconds each with a tennis ball, leaving a 20-second break between contractions. In the first set, the participant simply watched a video that showed a forearm performing the task, placed in the standard position and with the tennis ball in the hand. Once that first set was completed, the participant took a 2-minute break before starting the second set, in which they performed the 10 isometric contractions with the tennis ball while they watched the video.
  Interventions: Other: Mental Practise
- Control Group (Active Comparator): The participants in the control group were given instructions to perform a daily training of a single set. The set consisted of 10 isometric hand grip contractions for 3 seconds each with a tennis ball, leaving a 20-second break between contractions.
  Interventions: Other: Mental Practise

INTERVENTIONS:
Other: Mental Practise — They made a mental task to produce a neurophysiological activation of the brain areas related to the planning and execution of voluntary movement in a manner that resembles how the action is performed in reality in combination with real exercises.
  Other Names: Mental Task

SUMMARY:
Motor imagery is defined as a dynamic mental process of an action, without its real motor execution. Action observation training consists of watching an action performed by someone else. The primary objective of this study was to evaluate the effects of motor imagery and action observation combined with a hand grip strength program on strength gains in asymptomatic participants. The secondary objective was to assess the influence of motor imagery and action observation training combined with a hand grip strength program on electromyographic activity and intramuscular oxygenation of the forearm muscles.

DETAILED DESCRIPTION:
Motor imagery is defined as a dynamic mental process of an action, without its real motor execution. Action observation training consists of watching an action performed by someone else. Both motor imagery and action observation have been shown to produce a neurophysiological activation of the brain areas related to the planning and execution of voluntary movement in a manner that resembles how the action is performed in reality.

Several studies have shown that patients can report a significant improvement in strength with motor imagery training. There is also evidence regarding the improvements in motor skills in participants who perform motor imagery training combined with mirror therapy. Motor imagery is recognized as one of the most popular and effective forms of training to improve learning strategies and to increase the capacity to perfect sports movements, as has been observed in rhythmic gymnastics athletes.

In addition to the previously mentioned adaptations, a recent research proved that motor imagery and action observation provoke an activation of the sympathetic-excitatory nervous system. Changes in respiration, heart rate and skin temperature are produced, as well as an increase in electrodermal activity.

Both motor imagery and action observation are interventions that can generate adaptive neuroplastic changes on a cortical level, leading to a decrease in chronic pain. These rehabilitation techniques are used in pain treatment and impaired movement injuries that could be due to a nervous system alteration.

Action observation effectively facilitates motor learning, and is a tool for rehabilitation in neurological and musculoskeletal diseases. Action observation training leads to significant improvements in static balance and helps improve gait in patients with hemiparesis after an ictus.

A recent study showed that the patient's functionality loss is lessened if motor imagery and action observation are applied after an immobilization process, reducing the loss of wrist mobility, strength and muscle mass.

The effectiveness of motor imagery is controversial; several studies have presented unfavorable outcomes from this technique. Some variables, such as the duration of the sessions, the time employed the type of motor task or the number of sessions can influence the outcomes of these studies. Thus, it is necessary to clarify the controversial aspects of motor imagery, which lead us to perform this study.

This study evaluates variables that have not yet shown conclusive results: intramuscular oxygenation and electromyography. Focusing principally on the effectiveness of the treatment and the adaptations that are generated on an intramuscular level leads to a better understanding of what occurs as a result of training with motor imagery and action observation, and also whether these variables influence the effectiveness of the treatment.

Therefore, the primary objective of this study was to evaluate the effects of motor imagery and action observation combined with a hand grip strength program on strength gains in asymptomatic participants. The secondary objective was to assess the influence of motor imagery and action observation training combined with a hand grip strength program on electromyographic activity and intramuscular oxygenation of the forearm muscles.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic participants;
* men and women aged 18 to 65 years.

Exclusion Criteria:

* participants who had any knowledge of physical therapy;
* underage participants;
* participants with pain at the time of the study;
* participants with any type of neurological disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
The hand grip strength | Change in hand grip strength after 72 hours post-intervention
  The hand grip strength in kilograms was assessed using a Jamar dynamometer with the standard protocols for hand grip training. The measurements with the Jamar dynamometer present excellent test-retest reliability (intraclass correlation coefficient [ICC] = 0.81-0.99) for preferred and nonpreferred hands in men and excellent test-retest reliability (ICC = 0.83-1.0) for preferred and nonpreferred hands in women. The Jamar Dynamometer presents excellent intra-rater reliability (ICC = 0.94 and 0.98) and excellent inter-rater reliability (ICC = 0.98 for right and left handgrip strength).

SECONDARY OUTCOMES:
Intramuscular oxygenation | Change in Intramuscular oxygenation after 72 hours post-intervention
  The intramuscular oxygenation of the extensor muscles of the forearm was measured with the Moxy Monitor System. The Moxy sensor is placed over the muscle bellies of the extensor carpi radialis longus and the extensor carpi radialis brevis and measures the intramuscular oxygenation through a continuous infrared light emission.
Electromyographic activity | Change in Electromyographic activity after 72 hours post-intervention
  The electromyographic activity of the extensor muscles of the forearm was measured on the bellies of the extensor carpi radialis longus and the extensor carpi radialis brevis, placing the two electrodes in each of the muscle bellies, and a fifth electrode over the olecranon, which acts as a grounding. The Physioplux system was used for muscle contraction capture.

CONTACTS AND LOCATIONS:
Overall Officials: Roy A La Touche, PT, PhD, Study Director — Departamento de Fisioterapia. Centro Superior de Estudios Universitarios de La Salle. Universidad Autónoma de Madrid. Madrid. Spain
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No